CLINICAL TRIAL: NCT05249855
Title: Balneotherapy and Anxiety During SARS-CoV-2 Pandemic
Acronym: TRATACO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Bucharest (Other)
Responsible Party: Principal Investigator, Violeta Stefania Rotarescu, Researcher, University of Bucharest
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UBucharest
Record Dates: First submitted 2022-02-18; First posted 2022-02-22 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: D001452
Keywords: balneology; anxiety; fear of SARS-CoV-2; resilience; general trust
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: General Trust mediates the relation between the level of anxiety at the beginning of the treatment and the end of the treament.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Longitudinal Study (Other): A longitudinal study of anxiety over the balneological treatment.
  Interventions: Behavioral: Psychological measurement

INTERVENTIONS:
Behavioral: Psychological measurement — Psychological assessment

SUMMARY:
Investigators will measure the level of anxiety and fear of Covid during the balneological treatment in patients. They are interested in the effect of general trust and resilience on the level of anxiety state.

DETAILED DESCRIPTION:
Investigators will measure the level of anxiety and fear of SARS-CoV-2 virus during the balneological treatment in patients. They are interested in the effect of general trust and resilience on the level of anxiety state.

A number of between 300 and 800 inpatients are expected to get involved in the study. They suffer from cardiovascular disease, osteoarthritis, respiratory diseases and many others.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in balneological treatment

Exclusion Criteria:

* not enrolled in the balneological treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-05-20 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-11-15 (Estimated)

PRIMARY OUTCOMES:
Level of Anxiety | 10 days
  Low level of anxiety

IPD SHARING:
Plan to Share IPD: Undecided
The database will be uploaded to a database website.